CLINICAL TRIAL: NCT04112810
Title: A Phase II Trial of Tildrakizumab for Prevention of Acute Graft-Versus-Host Disease
Brief Title: Tildrakizumab for Prevention of Acute Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, William R. Drobyski, MD, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO35737
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Hematologic Malignancies
Keywords: Graft-versus-host disease
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease | interventions — tildrakizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tildrakizumab (Experimental): Tildrakizumab (IluymaTM) is a humanized monoclonal antibody that specifically binds to the IL-23p19 subunit of IL-23 to neutralize its function.
  Interventions: Drug: Tildrakizumab

INTERVENTIONS:
Drug: Tildrakizumab — 100 mg will be injected subcutaneously on Day -1, Day 28 ± 3, Day 112 ± 7, Day 196 ± 14, and Day 280 ± 14.
  Other Names: Iluyma

SUMMARY:
This is a phase 2 open-label trial designed to evaluate the efficacy of tildrakizumab in improving graft-versus-host disease (GVHD)-free relapse-free survival after myeloablative allogeneic hematopoietic cell transplantation (alloHCT) for hematologic malignancy.

DETAILED DESCRIPTION:
Study Rationale: GVHD remains a major cause of morbidity and mortality following myeloablative conditioning (MAC) alloHCT. Proinflammatory cytokines play a central role in initiation and development of acute GVHD and as such, inhibition of these cytokines has been examined for both prevention and treatment of GVHD. Interleukin (IL)-23 is a proinflammatory cytokine which the investigators' lab has shown to have a unique and selective role in induction of colonic inflammation during acute GVHD and that this cytokine serves as a critical mediator linking conditioning regimen-induced mucosal injury and endotoxin lipopolysaccharide (LPS) translocation to subsequent proinflammatory cytokine production and GVHD-associated pathological damage. Moreover, additional studies have demonstrated that blocking the IL-23 signaling pathway has not abrogated the graft-versus-tumor effect. Tildrakizumab is a commercially available anti-IL-23 antibody FDA approved for the treatment of moderate to severe psoriasis with good tolerance. The investigators hypothesize that blocking IL-23, with tildrakizumab, will reduce GVHD rates for patients undergoing MAC alloHCT without having an impact on relapse rates, thus improving GVHD-free relapse-free survival (GRFS).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Patients with any hematologic malignancy for which alloHCT is indicated. Patients with acute myeloid leukemia (AML) and acute lymphoblastic leukemia (ALL) must be in complete remission at the time of alloHCT (<5% blasts in the bone marrow, normal maturation of all cellular components in the bone marrow and absence of extramedullary disease). Patients with myelodysplastic syndrome (MDS) must have <10% blasts in the bone marrow, no circulating blasts.
3. Myeloablative conditioning (MAC) regimen, based on Center for International Blood and Marrow Transplant Research (CIBMTR) criteria (total body irradiation (TBI) ≥5 Gy single dose or ≥8 Gy fractionated or busulfan [Bu] dose >8 mg/kg oral or >6.4 mg/kg intravenous).
4. T cell-replete peripheral blood graft.
5. Patients must have a matched related or unrelated donor (at least 6/6 match at human leukocyte antigen (HLA) -A, -B and -C for related donors and at least 8/8 match at HLA -A, -B, -C and -DRB1 for unrelated donors).
6. Cardiac function: Left ventricular ejection fraction ≥45% for myeloablative conditioning.
7. Estimated creatinine clearance ≥40 mL/minute (using the Cockcroft-Gault formula and actual body weight).
8. Pulmonary function: diffusing capacity of the lungs for carbon monoxide (DLCO) ≥40% (adjusted for hemoglobin) and forced expiratory volume in 1 second (FEV1) ≥50%.
9. Liver function: total bilirubin <3 x upper limit of normal and alanine aminotransferase (ALT) / aspartate aminotransferase (AST) <5 x upper normal limit.
10. Female subjects must meet one of the following:

    Postmenopausal for at least one year before enrollment, OR
    1. Surgically sterile (i.e. undergone a hysterectomy or bilateral oophorectomy), OR
    2. If subject is of childbearing potential (defined as not satisfying either of the above two criteria), she must agree to practice two acceptable methods of contraception (combination methods require use of two of the following: diaphragm with spermicide, cervical cap with spermicide, contraceptive sponge, male or female condom, hormonal contraceptive) from the time of signing of the informed consent form through 90 days after the last dose of study agent, OR
    3. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods] and withdrawal are not acceptable contraception methods.)
11. Male subjects, even if surgically sterilized (i.e., status post vasectomy), must agree to one of the following:

    1. Practice effective barrier contraception during the entire study period and through 60 calendar days after the last dose of study agent, OR
    2. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post ovulation methods] and withdrawal are not acceptable methods of contraception.)
12. Signed informed consent: Voluntary written consent must be given before patient registration and performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
13. Planned post-transplant maintenance therapy is allowed.
14. Prior autologous transplant is allowed.

Exclusion Criteria:

1. Prior allogeneic hematopoietic cell transplant (HCT).
2. Active central nervous system (CNS) involvement with malignancy.
3. Patients receiving cord blood or haploidentical allograft.
4. Patients undergoing in vivo or ex vivo T cell-depleted alloHCT.
5. Karnofsky Performance Score <60% or Eastern Cooperative Oncology Group (ECOG) > or = 2.
6. Patients with uncontrolled bacterial, viral or fungal infections (currently on treatment and with progression of infectious disease or no clinical improvement) at time of enrollment.
7. Active hepatitis B or C virus infection or known human immunodeficiency virus (HIV) positive.
8. Use of rituximab, alemtuzumab, anti-thymocyte globulin (ATG) or other monoclonal antibody planned as part of conditioning regimen for GVHD prophylaxis.
9. Participation in another GVHD prophylaxis clinical trial.
10. Any current uncontrolled cardiovascular conditions, including uncontrolled ventricular arrhythmias, New York Heart Association (NYHA) class III or IV congestive heart failure, uncontrolled angina, or electrocardiographic evidence of active ischemia or active conduction system abnormalities.
11. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Drobyski, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Runaas L, Fank S, Palen K, Szabo A, Rein L, Ying G, Salzman N, Samanas L, Abedin SM, Chhabra S, Hamadani M, Longo W, Shah NN, Haber J, Gradissimo A, Waters NR, Peled JU, Johnson B, Kearl T, Drobyski WR. TIDRAKIZUMAB FOR THE PROPHYLAXIS OF GRAFT VERSUS HOST DISEASE AFTER ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION. Blood Adv. 2026 Feb 3:bloodadvances.2025019065. doi: 10.1182/bloodadvances.2025019065. Online ahead of print. PMID 41632629

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tildrakizumab
Started | 51
Completed | 50
Not Completed | 1
Not completed — Only 50 pts are evaluable as 1 pt withdrew before treatment. | 1

BASELINE CHARACTERISTICS:
Population: Fifty-one subjects enrolled. One subject withdrew before treatment. Technically, this patient should be included in the demographics table, because they were enrolled. However, since they received no study drug for non-study-related reasons, they are not part of either the safety population or the efficacy population.
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 47
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: GVHD-free Relapse-Free Survival
Description: Number of subjects experiencing any of grade III-IV acute GVHD, systemic therapy-requiring chronic GVHD, relapse, or death at 12 months
Time Frame: 1 year
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
percentage of subjects | 19.3 [11.8 to 31.4]

2. Secondary Outcome: Incidence of Chronic GVHD
Description: Number of subjects experiencing chronic GVHD defined by NIH Consensus criteria.
Time Frame: Day +180
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
percentage of subjects | 18 [10 to 32.5]

3. Secondary Outcome: Incidence of Chronic GVHD
Description: Number of subjects experiencing chronic GVHD defined by NIH Consensus criteria.
Time Frame: Day +365
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
percentage of subjects | 53.7 [40.4 to 68.9]

4. Secondary Outcome: Incidence of Acute GVHD
Description: Number of subjects experiencing grades II-IV and III-IV acute GVHD will be determined at Day +100 and Day +180 post-HCT. Acute GVHD will be graded according to NIH Consensus criteria.
Time Frame: Day +100 and Day +180
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
percentage of subjects
  Grade II-IV; Day +100 | 14 [7 to 27.8]
  Grade II-IV; Day +180 | 18 [10 to 32.5]
  Grade III-IV; Day +100 | 4 [1 to 15.6]
  Grade III-IV; Day +180 | 4 [1 to 15.6]

5. Secondary Outcome: Incidence of Acute GI GVHD
Description: Number of subjects experiencing grades II-IV and III-IV acute GI GVHD will be determined at Day +100 and Day +180 post-HCT. This will be graded according to NIH Consensus criteria.
Time Frame: Day +100 and Day +180
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
percentage of subjects
  Grade II-IV; Day +100 | 6 [2 to 18.1]
  Grade II-IV; Day +180 | 10.3 [4.5 to 23.7]
  Grade III-IV; Day +100 | 4 [1 to 15.6]
  Grade III-IV; Day +180 | 4 [1 to 15.6]

6. Secondary Outcome: Primary Graft Failure.
Description: Number of subjects experiencing no neutrophil recovery to > 500 cells/μL by Day 28 post-HCT.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
Participants | 0

7. Secondary Outcome: Secondary Graft Failure
Description: Number of subjects experiencing initial neutrophil engraftment followed by subsequent decline in absolute neutrophil counts <500 cells/μL, unresponsive to growth factor therapy, but cannot be explained by disease relapse or drugs.
Time Frame: Up to Day 365
Measure: Count of Participants; unit: Participants
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
Participants | 0

8. Secondary Outcome: Hematopoietic Recovery According to Neutrophil Count Recovery
Description: This measure is the number of subjects with the event. The number of days to hematopoietic recovery will be assessed according to neutrophil count recovery after hematopoietic stem cell transplant (HSCT). Neutrophil recovery or engraftment is defined as achieving an absolute neutrophil count (ANC) ≥500/mm^3 for three consecutive measurements on three different days. The first of the three days will be designated the day of neutrophil engraftment.
Time Frame: Day +28
Measure: Count of Participants; unit: Participants
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
Participants | 50

9. Secondary Outcome: Hematopoietic Recovery According to Platelet Count Recovery
Description: This measure is the number of subjects with the event. The number of days to hematopoietic recovery will be assessed according to platelet count recovery after HSCT. Platelet recovery is defined by either the first day of a sustained platelet count >20,000/mm^3 for three days with no platelet transfusion in the preceding seven days. The first day of sustained platelet count above these thresholds will be designated the day of platelet engraftment.
Time Frame: Day +28
Measure: Count of Participants; unit: Participants
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
Participants | 47

10. Secondary Outcome: Non-relapsed Mortality.
Description: Number of subjects who die after alloHCT without experiencing a relapse.
Time Frame: Day +100 and 1 year
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
percentage of subjects
  Day +100 | 2 [.3 to 13.9]
  1 year | 8 [3.1 to 20.5]

11. Secondary Outcome: Disease Relapse or Progression
Description: The number of subjects who experience relapse. Relapse is defined by either morphological, cytogenetic or radiologic evidence of the pretransplant hematologic malignancy.
Time Frame: Day +100 and 1 year
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
percentage of subjects
  Day +100 | 14 [7 to 27.8]
  1 year | 14 [7 to 27.8]

12. Secondary Outcome: The Number of Subjects With Progression-free Survival.
Description: This will be measured in months. The event for this endpoint is relapse/progression or death. Patients who are alive and disease-free will be censored at last follow-up.
Time Frame: Day +100 and 1 year
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
percentage of subjects
  Day +100 | 84 [74.4 to 94.8]
  1 year | 78 [67.3 to 90.4]

13. Secondary Outcome: The Number of Subjects With Overall Survival.
Description: The time in months from the date of transplant to date of death from any cause or for surviving patients, to last follow-up. Patients who are alive and disease-free will be censored at last follow-up.
Time Frame: Day +100 and 1 year
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
percentage of subjects
  Day +100 | 98 [94.2 to 100]
  1 year | 80 [69.7 to 91.9]

14. Secondary Outcome: Incidence of Infections
Description: Number of subjects experiencing a grade ≥3 (CTCAE v5) viral, fungal and/or bacterial infections.
Time Frame: Day +28, Day +100 and 1 year
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Tildrakizumab
Number analyzed (Participants) | 50
percentage of subjects
  Day +28 | 14 [7 to 27.8]
  Day +100 | 16 [8.5 to 30.2]
  1 Year | 20.3 [11.6 to 35.3]

ADVERSE EVENTS:
Time Frame: 12 months following alloHCT (up to 13 months)
Description: regular investigator assessment, regular laboratory testing
Arm/Group | Tildrakizumab
All-Cause Mortality (participants affected / at risk) | 10/50
Serious Adverse Events (participants affected / at risk) | 11/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tildrakizumab (N=50)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Blood bilirubin increased (Investigations) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Lung Infection - Lactobacillus (Infections and infestations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Embolisms (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Lung Infection (Infections and infestations) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Perineal Abscess (Reproductive system and breast disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tildrakizumab (N=50)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Acute kidney injuryAcute kidney injury (Renal and urinary disorders) | 4 (4)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 8 (11)
Anal pain (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 30 (79)
Anorexia (Metabolism and nutrition disorders) | 21 (26)
Anxiety (Psychiatric disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (6)
Aspartate aminotransferase increased (Investigations) | 6 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bladder perforation (Renal and urinary disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Microangiopathic Hemolytic Anemia (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (5)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 6 (7)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
non-productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Delirium (Psychiatric disorders) | 2 (3)
Dental caries (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 13 (17)
Dizziness (Nervous system disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (11)
Edema face (General disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 18 (24)
Febrile neutropenia (Blood and lymphatic system disorders) | 28 (30)
Fever (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Generalized edema (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2)
Veno-Occlusive Disease (VOD) (Hepatobiliary disorders) | 2 (2)
Herpes simplex reactivation (Infections and infestations) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 12 (17)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (16)
parainfluenza (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Skin GVHD (Investigations) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 4 (4)
Lymphocyte count decreased (Investigations) | 8 (16)
Mucositis oral (Gastrointestinal disorders) | 26 (31)
Nausea (Gastrointestinal disorders) | 13 (18)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neutrophil count decreased (Investigations) | 39 (116)
Non-cardiac chest pain (General disorders) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 7 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 42 (213)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Word finding difficulties (Psychiatric disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Catatonic (Psychiatric disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (16)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3)
COVID-19 Viral pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Sepsis (Infections and infestations) | 5 (5)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 17 (18)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Urethral infection (Infections and infestations) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal infection (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 40 (122)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT04112810/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT04112810/ICF_001.pdf